CLINICAL TRIAL: NCT00949117
Title: An Open Label Randomized Phase II Study of an Appetite Stimulant, Cyproheptadine Hydrochloride, With and Without a Nutritional Supplement, in Children With Cancer/Treatment-Related Weight Loss
Brief Title: Cyproheptadine Hydrochloride and Nutritional Supplementation in Treating Young Patients With Weight Loss With Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study not feasible with low accrual. DSMB recommended closure
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SCUSF 0802; SCUSF-0802 (Other: SunCoast CCOP Research Base); 5U10CA081920-11 (NIH)
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Leukemia; Lymphoma; Malnutrition; Myelodysplastic Syndromes; Unspecified Childhood Solid Tumor, Protocol Specific; Weight Changes
Keywords: malnutrition; weight changes; childhood acute lymphoblastic leukemia in remission; recurrent childhood acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia; childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; untreated childhood acute myeloid leukemia; other myeloid malignancies; stage I childhood Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood anaplastic large cell lymphoma; stage I childhood anaplastic large cell lymphoma; stage II childhood anaplastic large cell lymphoma; stage III childhood anaplastic large cell lymphoma; stage IV childhood anaplastic large cell lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; recurrent childhood large cell lymphoma; stage I childhood large cell lymphoma; stage II childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; childhood nasal type extranodal NK/T-cell lymphoma; childhood Burkitt lymphoma; recurrent childhood small noncleaved cell lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma; childhood myelodysplastic syndromes; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Leukemia; Lymphoma; Malnutrition; Myelodysplastic Syndromes; Body Weight Changes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Extranodal NK-T-Cell; Burkitt Lymphoma | interventions — Cyproheptadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I- cyproheptadine hydrochloride (Experimental): Patients receive oral cyproheptadine hydrochloride twice daily for up to 24 weeks in the absence of weight loss or unacceptable toxicity.
  Interventions: Drug: cyproheptadine hydrochloride
- cyproheptadine HCl & PediaSure or Ensure (Experimental): Patients receive oral cyproheptadine hydrochloride twice daily and oral PediaSure (2 to 10 years of age) or Ensure (> 10 years of age) twice daily for up to 24 weeks in the absence of weight loss or unacceptable toxicity.
  Interventions: Dietary Supplement: Ensure; Dietary Supplement: PediaSure; Drug: cyproheptadine hydrochloride

INTERVENTIONS:
Dietary Supplement: Ensure — Given orally
  Other Names: nutritional supplement drink
  Arms: cyproheptadine HCl & PediaSure or Ensure
Dietary Supplement: PediaSure — Given orally
  Other Names: nutritional supplement drink (pediatric)
  Arms: cyproheptadine HCl & PediaSure or Ensure
Drug: cyproheptadine hydrochloride — Given orally
  Other Names: cyproheptadine HCl

SUMMARY:
RATIONALE: Cyproheptadine hydrochloride may help improve appetite and lessen weight loss caused by cancer or cancer treatment. It is not yet known whether cyproheptadine hydrochloride is more effective with or without nutritional supplementation in improving weight and quality of life of young patients with weight loss caused by cancer or cancer treatment.

PURPOSE: This randomized phase II trial is studying cyproheptadine hydrochloride to see how well it works when given together with or without nutritional supplementation in treating young patients with weight loss caused by cancer or cancer treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the efficacy of an appetite stimulant, cyproheptadine hydrochloride, with vs without a nutritional supplement, PediaSure or Ensure, in improving weight and extending the duration of response in pediatric patients with cancer- or cancer treatment-related weight loss.

Secondary

* To compare patterns of body composition and weight change in patients treated with these regimens.
* To compare the change in the relationship between pre-albumin (biomarker of malnutrition) and weight improvement from baseline to the completion of study treatment.
* To compare the change in quality of life as measured by the Pediatric Functional Assessment of Anorexia and Cachexia Therapy (FAACT) questionnaire in patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center and steroid use (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral cyproheptadine hydrochloride twice daily for up to 24 weeks in the absence of weight loss or unacceptable toxicity.
* Arm II: Patients receive oral cyproheptadine hydrochloride twice daily and oral PediaSure (2 to 10 years of age) or Ensure (> 10 years of age) twice daily for up to 24 weeks in the absence of weight loss or unacceptable toxicity.

Patients undergo blood sample collection to assess pre-albumin levels at baseline and at weeks 4 and 24. Patients also undergo assessment of body composition, lean body mass, and percentage of body fat at baseline and at weeks 4 and 24 and assessment of weight and height at baseline and at weeks 4, 8, 12, 16, 20, and 24. Patients also complete a food diary twice a week during study treatment.

Patients 7-17 years of age complete a quality-of-life questionnaire at baseline and at weeks 4 and 24.

ELIGIBILITY:
INCLUSION CRITERIA:

* ≥ 2 years and < 18 years of age at the time of admission to the study
* Meets one of the following criteria:
* documented history of unintended weight loss > 5% presumed secondary to cancer/treatment-related therapy within three months
* BMI for age less than the 5th percentile
* Diagnosed with cancer of any type
* Concomitant cancer treatment (surgery, chemotherapy, radiotherapy) guidelines:
* Patients who will complete concomitant cancer treatment during this study's 4-week intervention are not eligible
* If patients are receiving concomitant cancer treatment, they should be scheduled to get at least another 4 weeks of treatment in order to reach the primary endpoint
* If patients have already completed cancer treatment, they need to be enrolled within 8 weeks of completing therapy.
* Predicted life expectancy of at least 6 months

EXCLUSION CRITERIA:

* Currently taking any of the study agents (cyproheptadine hydrochloride (CH), PediaSure, or Ensure) or have taken any of the study agents during the past 3 weeks
* History of anorexia nervosa or bulimia
* Initiation of other appetite enhancing agents including steroids prescribed for the intent of weight gain, i.e. Megace, is not allowed during this study
* Children receiving steroids as part of their daily cancer treatment regimen are excluded from participation. However, intermittent steroid use in an antiemetic regimen or in other pulse steroid therapy is allowed during the study.
* Use of other forms of nutrition therapies, e.g. total parenteral nutrition (TPN) or enteral tube feedings within 3 weeks of study entry or during study
* Receiving monoamine oxidase (MAO) inhibitors, procarbazine, fluoxetine (SSRI), or paroxetine (SSRI)
* Taking dronabinol (Marinol) or other appetite-stimulating medications during the past 3 weeks
* Diagnosed with glaucoma, cystic fibrosis, inflammatory bowel disease or GI or genitourinary (GU) obstruction
* Allergy to study agents
* Hypersensitivity to specific milk proteins
* Pregnant or lactating. Females of childbearing potential are required to use effective contraception while on study agent.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Couluris, DO, Study Chair — University of South Florida

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm II Cyproheptadine HCl and PediaSure or Ensure: Patients receive oral cyproheptadine hydrochloride twice daily and oral PediaSure (2 to 10 years of age) or Ensure (> 10 years of age) twice daily for up to 24 weeks in the absence of weight loss or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I- Cyproheptadine Hydrochloride | Arm II Cyproheptadine HCl and PediaSure or Ensure
Started | 4 | 5
Completed | 1 | 0
Not Completed | 3 | 5
Not completed — Lack of Efficacy | 2 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I- Cyproheptadine Hydrochloride | Arm II Cyproheptadine HCl and PediaSure or Ensure | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 9
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (5.5) | 13.3 (5.1) | 11.4 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Measures of Weight at Baseline and at Week 24
Description: Difference in measure of weight in kilograms of subject at baseline and at week 24 after continuing on study treatment for the entire 24 week period.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Arm I- Cyproheptadine Hydrochloride | Arm II Cyproheptadine HCl and PediaSure or Ensure
Number analyzed (Participants) | 1 | 0
kilograms | 4.3 |

2. Secondary Outcome: Body Mass Index as Assessed at Baseline and 24 Weeks
Description: Change in Body Mass Index (BMI) in subjects from Baseline visit to 24 week visit.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Arm I- Cyproheptadine Hydrochloride | Arm II Cyproheptadine HCl and PediaSure or Ensure
Number analyzed (Participants) | 1 | 0
kg/m^2 | 1.9 |

3. Secondary Outcome: Effect of Cyproheptadine Hydrochloride on Pre-albumin and Body Composition
Time Frame: 24 weeks
Population: Outcome not assessed as the one subject that completed the protocol did not have the prealbumin lab drawn at the 24 week visit and body composition tests assessed.
Arm/Group | Arm I- Cyproheptadine Hydrochloride | Arm II Cyproheptadine HCl and PediaSure or Ensure
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Quality of Life as Assessed by Peds-FAACT Questionnaire at Baseline and at Weeks 4 and 24
Time Frame: 24 weeks
Population: Outcome not assessed as the one subject that completed the protocol was too young to complete the PedsFAACT quality of life assessment.
Arm/Group | Arm I- Cyproheptadine Hydrochloride | Arm II Cyproheptadine HCl and PediaSure or Ensure
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Weight for Age Z-score From Baseline Through 24 Weeks
Description: Change in weight for age Z-score from Baseline through 24 weeks while on study treatment. Weight for age Z-score calculated using the Center for Disease Control and Prevention (CDC) weight-for-age Z score data tables.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Arm I- Cyproheptadine Hydrochloride | Cyproheptadine HCl & PediaSure or Ensure
Number analyzed (Participants) | 1 | 0
z score | 1.47 (0) |

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Subjects and their parents reported any adverse symptoms or events via daily study medication logs. Site personnel reviewed logs at in-person visits at weeks 4, 8, 12, 16, 20 and 24 and assessed subject for any adverse events. All Adverse events and Serious Adverse events reviewed by independent DSMB.
Arm/Group | Arm I- Cyproheptadine Hydrochloride | Arm II Cyproheptadine HCl and PediaSure or Ensure
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 1/4 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I- Cyproheptadine Hydrochloride (N=4) | Arm II Cyproheptadine HCl and PediaSure or Ensure (N=5)
somnolence (General disorders) | 1 (1) | 0 (0)
relapse of cancer (General disorders) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study closed early due to slow accrual and lack of feasibility Only 1 subject completed protocol and considered in the outcome measures. Subject too young to complete PedsFAACT & did not have prealbumin drawn at 24 week visit so outcomes not assessed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No